CLINICAL TRIAL: NCT04767568
Title: Exploratory Study of the Relevance of a Blood Test in the Management of Patients in the Context of Colorectal Cancer Screening
Acronym: PREDICT-IRFC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/539
Record Dates: First submitted 2020-12-03; First posted 2021-02-23 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer
Keywords: blood test; early detection
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood test (Experimental): In Cohort A: 200 patients with suspected colorectal cancer following a positive immunological test during screening (presence of blood detected in the stool) OR with gross bleeding
  In cohort B: 200 patients who have already performed colonoscopy candidates for surgery on their colorectal tumor
  Interventions: Diagnostic Test: Blood sample; Other: Tumor tissue; Other: stool collection

INTERVENTIONS:
Diagnostic Test: Blood sample — In cohort A: Blood sample n°1 (PBMC, plasma, ctDNA) previous colonoscopy. If no cancer lesions: STOP. If cancer lesion detected : Blood sample n°2 (PBMC, plasma, ctDNA) collected 1 month after surgery.
  In cohort B: Blood sample n°1 (PBMC, plasma, ctDNA) collected before surgery. Blood sample n°2 (PBMC, plasma, ctDNA) collected 1 month after surgery
Other: Tumor tissue — In each cohort, tumor tissue will be collected from the surgical specimen.
Other: stool collection — In cohort B: Stool sample n°1 collected before surgery. Stool sample n°2 collected 1 month after surgery

SUMMARY:
Colorectal cancer (CRC) is the third most common cancer in men and the second in women with an incidence of 43,350 new cases in 2018. This incidence is increasing every year.

Early detection is crucial in this pathology. In France, free screening is organized by health insurance for people aged 50 to 74 years. This screening is based on an immunological test (FIT: Fecal Immunological test), which aims to detect the presence of blood in the stool. In fact, some polyps or cancers cause bleeding that is often minimal and therefore difficult or even impossible to detect with the naked eye.

If this test is positive, a colonoscopy is done to check whether or not abnormalities are present in the colon or rectum. Performed under anesthesia, this examination can detect the possible presence of polyps or cancer.

Recently, with the covid-19 epidemic, the investigators were faced with an extension of the delays for colonoscopies which led to delays in patient care.

To prevent this, they propose to develop a blood test that would allow rapid identification of patients with colorectal cancer, requiring rapid management.

This blood test will permit to have a parameter for stratifying the therapeutic care in the event of epidemia or situation that constrains the organisation of the health system.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than18 years
* Cohort A : patients with suspected colorectal cancer following a positive immunological test during screening (presence of blood detected in the stool) or with gross bleeding OR Cohort B : patients who have already performed colonoscopy (on symptoms, or because of family history, or other ...), for whom the diagnosis of adenocarcinoma was identified by pathology prior to surgery, candidates for surgery on their colorectal tumor
* Signed and dated informed consent
* Patient affiliated to or beneficiary of French social security system.

Exclusion Criteria:

* Vulnerable persons according to the law (minors, adults under protection, persons deprived of liberty ...)
* Not ability to comply with the study protocol, in the Investigator's judgment
* pregnant woman
* Patient in the period of exclusion of another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of a blood test | one month after surgery, an average of 6 months from inclusion
correlation between the biological signature of the test and the stage of the disease in patients whose diagnosis of adenocarcinoma was identified by pathology prior to surgery. | one month after surgery, an average of 6 months from inclusion

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Besançon, Besançon
  - Hôpital Nord-Franche-Comté, Montbéliard
  - Centre Hospitalier Intercommunal de Haute-Saône, Vesoul